CLINICAL TRIAL: NCT01278641
Title: Men With Fibromyalgia or Chronic Widespread Pain - Effect of Exercise on Symptoms and Body Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Kaisa Mannerkorpi, Associate professor, Göteborg University, Dep of Rheumatology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 082-07
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2008-04

CONDITIONS: Fibromyalgia; Pain
Keywords: Fibromyalgia; Widespread pain; Fatigue; Physical exercise
MeSH Terms: conditions — Fibromyalgia; Pain; Fatigue; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Intervention i arm 1 comprises graded strength resistance training, 75 minutes twice a week for 12 weeks.
  Interventions: Behavioral: Graded strength resistance training program
- 2 (Experimental): Intervention in arm 2 comprises low intensive temperate pool exercise 50 minutes, twice a week for 12 weeks.
  Interventions: Behavioral: Temperate pool exercise program
- 3 (No Intervention): Reference group, continues with normal activities during the study period of 12 weeks.

INTERVENTIONS:
Behavioral: Graded strength resistance training program — Graded strength resistance training, 75 minutes, twice a week for 12 weeks.
  Arms: 1
Behavioral: Temperate pool exercise program — Temperate pool low intensive exercise, 50 minutes, twice a week for 12 weeks.
  Arms: 2

SUMMARY:
A controlled randomised trial (CRT). 60 men who fulfil the ACR-criteria for Fibromyalgia or Chronic Widespread Pain (Wolfe 1990) participate in the study.

The main objective of the study is to compare the effect of a graded strength training program and a low intensive pool exercise program.

DETAILED DESCRIPTION:
A controlled randomised trial (CRT). 60 men who fulfil the ACR-criteria for Fibromyalgia or Chronic Widespread Pain (Wolfe 1990) participate in the study.

40 patients (in the city Uddevalla) are randomised into two groups; low intensive temperate pool exercise program, and graded strength training program. The study period is 12 weeks.

20 patients (in the city Alingsås) make a reference group who is asked to continue their normal activities during the study period.

Primary outcomes are fatigue (using the Multidimensional fatigue inventory and VAS for global fatigue)and muscle strength (using Steve Strong, Isobex and the Grippit). Several other self-administered instruments was used.

ELIGIBILITY:
Inclusion Criteria:

Male patients with Fibromyalgia or Chronic Widespread pain

Exclusion Criteria:

Other severe physical or psychiatric disorders.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2008-01; Primary Completion 2009-03 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
The multidimensional Fatigue Inventory (MFI-20) | 12 weeks

SECONDARY OUTCOMES:
The Hospital Anxiety and Depression Scale (HADS) | 12 weeks
Muscle strength (measured with Isobex and Steve Strong) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kaisa E Mannerkorpi, Ass Prof, Principal Investigator — Göteborg University, Dept of Rheumatology
Locations (1):
- Sjukgymnastik Primärvård Rosenhäll, Uddevalla, Sweden

REFERENCES:
- [Derived] Ericsson A, Bremell T, Cider A, Mannerkorpi K. Effects of exercise on fatigue and physical capacity in men with chronic widespread pain - a pilot study. BMC Sports Sci Med Rehabil. 2016 Sep 6;8(1):29. doi: 10.1186/s13102-016-0054-9. eCollection 2016. PMID 27602228